CLINICAL TRIAL: NCT01948102
Title: Identification of Diagnostic and Prognostic Biomarkers From Amyotrophic Lateral Sclerosis (ALS) Skin and Adipose Samples
Acronym: ALS-TDI PEG
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: ALS Therapy Development Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CHS-Neurology_ALS_TDI_PEG
Record Dates: First submitted 2013-03-30; First posted 2013-09-23 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2019-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; motor neuron disease; biological markers; biomarkers
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin and adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- subjects with ALS: subjects with ALS who are undergoing a percutaneous endoscopic gastrostomy
- subjects without ALS: subjects without ALS who are undergoing a percutaneous endoscopic gastrostomy

SUMMARY:
The purpose of the project is to obtain skin and adipose tissue samples from patients with ALS to develop new diagnostic and prognostic markers of the disease. These samples will be obtained when percutaneous endoscopic gastrostomy (PEG) is performed as part of their standard of care. Skin and adipose tissue samples will also be obtained from disease control subjects who require a PEG as part of their standard of care.

DETAILED DESCRIPTION:
Subjects who are undergoing a percutaneous endoscopic gastrostomy (PEG) tube insertion as part of their standard of care will be asked if a skin and adipose sample may be collected for research during the procedure. After a participant has signed the informed consent, the sub-investigator from the Department of Gastroenterology will collect a skin and adipose sample during the procedure. Individuals with a diagnosis of definite ALS and disease controls (i.e. stroke, head and neck cancer, spinal cord injury, etc.) will be included in this study.

The coded skin and adipose sample will be taken to the Carolinas Neuromuscular/ALS Research Laboratory in the Cannon Research Center for processing. The skin and adipose will be separated from each other and divided into halves. Each half of skin and adipose will be submerged in preservative and either shipped to ALS-TDI or retained at -80°C in the Carolinas Neuromuscular/ALS Research Laboratory. The research staff at the Carolinas Neuromuscular/ALS-MDA Center will be responsible for shipping the sample to the ALS-TDI for either RNA isolation using the Qiagen RNAEasy kit (Qiagen) or for purification of protein. Subsequently, gene expression profiling on Affymetrix Genechips or Mass Spec based proteomics on a Thermo Orbitrap LC-MS/MS instrument will be performed, respectively. The discovery effort (if all participants are working at capacity) should not take more than 12 months.

In addition to the above procedures, a member of the study team will review the medical chart to obtain additional information on the participant's medical and family history. For ALS patients, past ALSFRS-R scores or FVC scores will be provided to the "ALS-TDI Skin and Adipose Biomarker Study" to enhance the usefulness of the information for research.

Samples will not be stored with any patient identifiers. Samples will be retained and continued to be studied as new techniques become available. Data from the study may be published in scientific journals. Publications will not include any patient identifiers.

ELIGIBILITY:
Inclusion Criteria:

* for ALS patients, subjects must be diagnosed with definite ALS according to the El Escorial Criteria (EEC)
* all subjects must be diagnosed with a condition requiring PEG (percutaneous endoscopic gastrostomy) tube insertion
* subjects must be older than 18 years of age

Exclusion Criteria:

* children 18 years old and younger

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the Carolinas Neuromuscular/ALS-MDA Center and patients at Carolinas Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2008-08-20 (Actual); Primary Completion 2014-08-06 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Abundance levels of the known messenger RNA transcriptome of skin and adipose tissue samples (measured by gene expression profiling) | After tissue has been collected from study subjects. Data will be analyzed at 1 year.
  Skin and adipose samples will be collected and processed into total RNA. Probes will be synthesized from these total RNAs and hybridized to HgU133ver2.0 Affymetrix genechips. These genechips contain probe sets that measure the abundance levels of the known human transcriptome.
Changes in abundance of or post-translational modification of proteins (measured by proteomics) | After tissue has been collected from study subjects. Data will be analyzed at year 1 after primary outcome data has been reviewed and analyzed.
  Skin and adipose samples will be collected for down stream proteomics analysis. The 14 most abundant proteins will be removed using commercially available depletion columns (Agilent). Removal of these proteins yields higher resolution and sensitivity in subsequent chromatography steps. Proteins will be separated by 2 and 3 dimensional liquid chromatography followed by MS/MS based peptide quantitation and sequencing on a Thermo Orbitrap.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin R Brooks, MD, Principal Investigator — Carolinas Neuromuscular/ALS-MDA Care Center; Thomas Pacicco, MD, Principal Investigator — Gastroenterology
Locations (1):
- Carolinas Neuromuscular/ALS-MDA care Center, Charlotte, North Carolina, United States